CLINICAL TRIAL: NCT04741893
Title: Assessment of the Effect of Ageing on Anal Sphincter Distensibility in Hong Kong Using EndoFLIP
Brief Title: Anal Canal Functional Assessment Using EndoFLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kaori Futaba, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CREC2017.125
Record Dates: First submitted 2018-02-19; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Faecal Incontinence; Asymptomatic Condition
Keywords: Faecal incontinence; Functional Lumen Imaging Probe; Anal distensibility
MeSH Terms: conditions — Encopresis; Asymptomatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- faecally incontinent patients (Experimental): faecally incontinent patients are all assessed using EndoFLIP as well as anorectal manometry and endoanal ultrasound
  Interventions: Device: EndoFLIP
- Asymptomatic individuals (Experimental): asymptomatic individuals are all assessed using EndoFLIP as well as anorectal manometry and endoanal ultrasound
  Interventions: Device: EndoFLIP

INTERVENTIONS:
Device: EndoFLIP — Use of Endoluminal Functional Lumen Imaging Probe to assess anal canal function

SUMMARY:
Faecal incontinence (FI) is characterized by involuntary loss of rectal content through the anal canal. FI is psychologically and socially debilitating problem that can dramatically affect patient's quality of life, often in otherwise healthy individual. FI can occur as a result of obstetric sphincter injury, surgery, irradiation, anorectal malformations as well as neurological, connective tissue or endocrine disorders. Currently management options for these patients are limited, partly due to the fact that control of defaecation and continence is multifactorial but also due to the fact that FI is difficult to identify the exact cause of patients' incontinence.

Current assessment of patients with FI include endoscopic assessment to rule out intraluminal organic cause for patients' symptoms, endoanal ultrasound scan / MRI to assess their pelvic floor anatomy and anorectal manometry to assess anorectal function. Anorectal manometry is a simple test to perform but Anorectal manometry is susceptible to measurement artifacts, with a high inter-individual variation with significant overlap between healthy asymptomatic and symptomatic patients with FI. Harris et al in 1966 suggested that the anal sphincter's resistance to distension that may be of importance for sphincter competence, not how tight anal sphincter can squeeze.

Endoluminal Functional Lumen Imaging Probe (EndoFLIP©) is a novel technology used to measure the dimensions and function of a hollow organ. Limited publication so far has shown that EndoFLIP© provides a new way of assessing anal sphincter competence. The study is to assess the use of EndoFLIP© to assess anal sphincter function in Hong Kong population. Firstly to evaluate whether age has an effect on the distensibility of the anal sphincter and its function and secondly to compare between symptomatic patients with faecal incontinence and asymptomatic healthy subjects.

ELIGIBILITY:
For Asymptomatic Group:

Inclusion Criteria: adults over 30 with no history of faecal incontinence, who are able to give consent.

Exclusion Criteria: Patients with history of gastrointestinal disease on medication or neurological disorder with bowel symptoms, anorectal surgery or previous bowel resection. Patients who are not willing to undergo the specified tests in this study. Pregnant women.

For Faecally Incontinent Group:

Inclusion Criteria: Adults over 30 with history of faecal incontinence for over 3months, who are able to give consent.

Exclusion Criteria: Patients who are not willing to undergo the specified tests in this study. Pregnant women and patients who has had anorectal surgery or bowel resection.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Change in anal distensibility with age in asymptomatic individuals assessed with EndoFLIP | 1 day
  Comparison of anal distensibility in between different age groups in asymptomatic individuals
Abnormal anal distensibility in faecally incontinent group | 1 day
  Comparison of anal distensibility between faecally incontinent patients and asymptomatic individuals using EndoFLIP

CONTACTS AND LOCATIONS:
Overall Officials: Kaori Futaba, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Harris LD, Winans CS, Pope CE 2nd. Determination of yield pressures: a method for measuring anal sphincter competence. Gastroenterology. 1966 Jun;50(6):754-60. PMID 5212375
- [Background] Sorensen G, Liao D, Lundby L, Fynne L, Buntzen S, Gregersen H, Laurberg S, Krogh K. Distensibility of the anal canal in patients with idiopathic fecal incontinence: a study with the Functional Lumen Imaging Probe. Neurogastroenterol Motil. 2014 Feb;26(2):255-63. doi: 10.1111/nmo.12258. Epub 2013 Nov 29. PMID 24286561
- [Background] Gourcerol G, Granier S, Bridoux V, Menard JF, Ducrotte P, Leroi AM. Do endoflip assessments of anal sphincter distensibility provide more information on patients with fecal incontinence than high-resolution anal manometry? Neurogastroenterol Motil. 2016 Mar;28(3):399-409. doi: 10.1111/nmo.12740. Epub 2015 Dec 15. PMID 26670599